CLINICAL TRIAL: NCT06769269
Title: Hypertension Registry: Study of Primary and Secondary Hypertension Phenotypes, Complications, and Treatment Personalization.
Status: Recruiting | Type: Observational
Sponsor: Moroccan Society of Cardiology (Other)
Collaborators: F&C Clinical Trials (Unknown)
Responsible Party: Sponsor
Other Study IDs: MoroccanSocietyCardiology
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The quality of primary healthcare systems for patients with hypertension (HTA) in Morocco is a critical issue due to its high prevalence and significant impact on morbidity and mortality. The concept of "quality in primary care" encompasses fundamental aspects such as timeliness, accessibility, and the provision of care based on current clinical guidelines and recommendations from professional societies.

This observational study on hypertension (HTA) uses an electronic registry accessible remotely to collect medical data from primary care and hospital settings. Investigators will be trained to ensure standardization in blood pressure measurements to minimize errors. The registry will include clinical, therapeutic, and complication data for patients aged 18 and over with a confirmed diagnosis of HTA, with information transmitted anonymously via a certified secure channel.

Informed consent from patients will be required for including their data in the registry. Collected data will include anthropometric measurements (weight, height, waist circumference, body mass index), blood pressure measurements by validated devices or ambulatory measurements, and metabolic assessments (blood glucose, total cholesterol, triglycerides, LDL, HDL, urea, creatinine, uric acid, urine albumin-to-creatinine ratio). Cardiovascular complications will also be recorded.

The study design is a cohort study with a cross-sectional perspective and a targeted follow-up period of one year. The study aims to evaluate the prevalence and phenotypes of HTA in Morocco, as well as the geographic distribution of the disease. It will compare current data with those from previous years and other North African countries to assess the applicability of Moroccan clinical practices and recommendations from the European Society of Cardiology (ESC). The goal is to enhance the understanding and management of HTA, as well as to optimize prevention and treatment strategies.

This comprehensive analysis will help identify potential gaps in primary care and develop strategies to improve the management of hypertensive patients. The comparative evaluation of data related to examinations, treatments, and complications of the cohort of patients followed for hypertension during the period 2024-2026, in comparison with results from previous years and other countries, will provide valuable insights into the shortcomings and progress in care delivery. This approach will not only identify areas needing improvement but also highlight significant advances in hypertension management.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged over 18 years.
* Patients with blood pressure:

  * Higher than 140 mmHg systolic and/or higher or equal to 90 mmHg diastolic in consultation or in a hospital setting.
  * Higher than 135/85 mmHg at home or in ambulatory blood pressure measurements (ABPM).
* Patients who have agreed and signed the informed consent.
* Patients with legal status in the Moroccan kingdom.

Exclusion Criteria:

* Patient without diagnosis of hypertension
* Patient under 18 years old
* Patients refusing to sign the informed consent.
* Patients with illegal status in the kingdom.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from various public and private research centers, whether they are already under follow-up for hypertension or newly diagnosed. Various specialists will be involved in the registry to increase the diversity of recruited patients, including cardiologists, general practitioners, and nephrologists. The objective is also to identify best practices for managing hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2027-01-21 (Estimated)

PRIMARY OUTCOMES:
Prevalence of arterial hypertension | At inclusion
  Proportion of population with arterial hypertension in Morocco.
To assess the distribution of HTA across the kingdom | At inclusion
  Analyzing how arterial hypertension is spread geographically and demographically within the kingdom.
To analyze the various phenotypes of primary and secondary hypertension as well as the associated complications | At inclusion
  Studying the different forms or presentations of hypertension (both primary and secondary) and their related health impacts, such as organ damage or cardiovascular events.
Causal relationships between Arterial Hypertension and various complications | At inclusion
  Causal relationships between arterial hypertension and various complications such as myocardial infarction, heart failure, atrial fibrillation, renal failure, and stroke, as well as links between arterial hypertension and other secondary pathologies

SECONDARY OUTCOMES:
Collect information on complications related to arterial hypertension after 1 year | 1 year

CONTACTS AND LOCATIONS:
Locations (5):
- Morocco (5):
  - Moroccan Society of Cardiology, Meknes, Morocco
  - Moroccan Society of Cardiology, Casablanca
  - UM6SSP, Casablanca
  - Ibn Sina Hospital Center, Rabat
  - Mohamed V Military Hospital, Rabat

IPD SHARING:
Plan to Share IPD: No